CLINICAL TRIAL: NCT05715853
Title: Prospective Assessment of Rejection in Kidney Transplant (PARK)
Acronym: PARK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: NephroSant (Industry)
Responsible Party: Sponsor
Other Study IDs: NEPHRO-002
Record Dates: First submitted 2023-01-27; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Kidney Transplant Failure and Rejection
Keywords: kidney transplant; kidney biopsy; allograft rejection
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: QSant — QSant™ is a needle free urine test collected in-home or in-clinic to aid in the evaluation and management of kidney transplant recipients' allograft status. QSant evaluates 6 kidney-specific biomarkers.

SUMMARY:
The PARK study is a multi-center observational study to assess the performance of the QSant test with kidney biopsy.

QSant is a test based on 6 urinary biomarkers that is used for the evaluation and management of acute rejection in renal allograft recipients with clinical suspicion of rejection.

DETAILED DESCRIPTION:
Non-randomized, unblinded observational study to collect urine samples, coincident allograft biopsy results, and relevant clinical data to evaluate the QSant test.

Participants will be recruited prior to or on the day of an already scheduled kidney biopsy.

Urine samples will be collected before biopsy (protocol and for-cause).

ELIGIBILITY:
Inclusion Criteria:

1. Kidney transplant recipient ≥ 18 years who are scheduled for kidney biopsy.
2. Kidney biopsy scheduled on a date > 14 days post-transplant
3. Able to understand risks and requirements of participation and provide informed consent
4. Willing and able to comply with the study requirements

Exclusion Criteria:

1. Inability to provide a voided urine sample per collection protocol
2. Urological abnormalities such as catheters, augmented bladder, ileal conduits, mitrofanoff, and vesicostomy
3. History of or current multi-organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult kidney transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Collect coincident urine specimens and biopsy results from participants | Prior to biopsy
  Collect urine sample using QSant kit for adult kidney transplant recipients
QScore specificity and sensitivity in relation to kidney biopsy | Prior to biopsy
  Evaluate the QSant algorithm performance in terms of sensitivity, specificity, and accuracy

CONTACTS AND LOCATIONS:
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States